CLINICAL TRIAL: NCT03129867
Title: Incidence and Models of Ticagrelor Discontinuation in Patients With Acute Coronary Syndrome
Brief Title: ADHerence of ticagrelOr in Real World Patients With aCute Coronary Syndrome
Acronym: AD-HOC
Status: Completed | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: AD-HOC
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 60mg or 90 mg as routine use of each Center
  Other Names: Brilique

SUMMARY:
Ticagrelor 90 mg twice daily treatment is recommended for 12 months in patients with acute coronary syndrome (ACS) and in patients undergoing coronary revascularization and conservative strategies. Recent data from the PEGASUS-TIMI 541 trial have shown that long-term treatment with ticagrelor reduced the risk of major cardiovascular adverse events (MACE) in stable ambulatory patients with a history of myocardial infarction. Based on these data, prolongation over 12 months of ticagrelor therapy could be indicated in selected patients; even if with such a prolongation some adverse effects on the treatment could be observed. In the PLATO2 trial, where median duration of exposure to the study drug was 277 days, the suspension of ticagrelor therapy was 7.4% in ticagrelor versus 6% in patients receiving clopidogrel ( P <0.001). Ticagrelor treatment interruption was mainly driven by non-serious adverse events occurring mainly shortly after randomization. For patients after the first year of treatment, the subsequent rate of interruption was low. These data demonstrate that adverse events considered "not serious" by traditional trial criteria may have an effect on quality of life and, therefore, can cause treatment interruption; The phenomenon emphasizes at the same time the importance of patient education and advice on timing and the nature of adverse effects in order to improve adherence. Patients in the real world may show a premature suspension rate of the drug even higher than in clinical trials. However, data from real-world patients is scarce.

DETAILED DESCRIPTION:
Ticagrelor 90 mg twice daily treatment is recommended for 12 months in patients with acute coronary syndrome (ACS) and in patients undergoing coronary revascularization and conservative strategies. Prolongation over 12 months of ticagrelor therapy could be indicated in selected patients; even if with such a prolongation some adverse effects on the treatment could be observed. In the PLATO2 trial, where median duration of exposure to the study drug was 277 days, the suspension of ticagrelor therapy was 7.4% in ticagrelor versus 6% in patients receiving clopidogrel ( P <0.001). Ticagrelor treatment interruption was mainly driven by non-serious adverse events occurring mainly shortly after randomization. For patients after the first year of treatment, the subsequent rate of interruption was low. These data demonstrate that adverse events considered "not serious" by traditional trial criteria may have an effect on quality of life and, therefore, can cause treatment interruption; The phenomenon emphasizes at the same time the importance of patient education and advice on timing and the nature of adverse effects in order to improve adherence. Patients in the real world may show a premature suspension rate of the drug even higher than in clinical trials. However, data from real-world patients is scarce.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>=18 years age) patients
* Patients discharged from the hospital with a diagnosis of ACS
* Patients discharged on ticagrelor therapy
* Patients who have signed an informed consent to study participation

Exclusion Criteria:

* Patients taking part in a study with a medical device or experimental drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients discharged from the hospital with a diagnosis of ACS and on ticagrelor therapy
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of drug discontinuation | At 12 months
  Ticagrelor discontinuation procedures include discontinuation, interruption and disruption. Discontinuation is defined as the definitive suspension recommended by physician for patients who are believed to no longer need ticagrelor. Interruption is defined as the temporary cessation of antiplatelet therapy for surgical needs with ticagrelor resumption after surgery. Disruption of therapy includes cessation of antiplatelet treatment due to bleeding or non-compliance

SECONDARY OUTCOMES:
Incidence of major adverse cardiac events (MACE) | At 12 months
  Incidence of major adverse cardiac events (MACE)
Incidence of major bleeding | At 12 months
  Incidence of major bleeding
Incidence of drug discontinuation | At 24 months
  Incidence of drug discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Fiocca, MD, Principal Investigator — ASST Papa Giovanni XXIII

IPD SHARING:
Plan to Share IPD: No